CLINICAL TRIAL: NCT06245291
Title: A Phase 2a, Open-Label Multiple Dose Study Evaluating the Safety, Tolerability, and Pharmacodynamics of Imdusiran (AB-729) in Combination With Intermittent Dosing of Durvalumab, a PD-L1 Monoclonal Antibody, in Subjects With Chronic HBV Infection
Brief Title: Study of Imdusiran (AB-729) in Combination With Intermittent Dosing of Durvalumab in Subjects With Chronic HBV Infection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Arbutus Biopharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB-729-203
Record Dates: First submitted 2024-01-11; First posted 2024-02-07 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort A (Experimental): Imdusiran 60 mg SC Q8 weeks + nucleos(t)ide analog for 48 weeks + durvalumab at early and mid-treatment period timepoints
  Interventions: Drug: Imdusiran; Drug: Durvalumab
- Cohort B (Experimental): Imdusiran 60 mg SC Q8 weeks + nucleos(t)ide analog for 48 weeks + durvalumab at mid and late-treatment period timepoints
  Interventions: Drug: Imdusiran; Drug: Durvalumab
- Cohort C (Experimental): Imdusiran 60 mg SC Q8 weeks + nucleos(t)ide analog for 48 weeks + durvalumab at 2 late treatment period timepoints
  Interventions: Drug: Imdusiran; Drug: Durvalumab

INTERVENTIONS:
Drug: Imdusiran — subcutaneous injection
Drug: Durvalumab — intravenous injection

SUMMARY:
This is a phase 2a, open-label, multicenter study investigating the safety, tolerability, and antiviral activity of durvalumab administered at targeted times during a 48-week treatment period of imdusiran in virologically-suppressed CHB subjects

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female between the ages of 18-65
* Willing and able to provide informed consent
* Willing to follow protocol-specified contraception requirement

Key Exclusion Criteria:

* Have extensive fibrosis or cirrhosis of the liver
* Have or had liver cancer (hepatocellular carcinoma)
* Family history or personal history/current thyroid disease on or off replacement therapy
* Have a history or current autoimmune disease or has been on immunosuppressive medications within 6 months of the start of the study
* Females who are breastfeeding, pregnant or who wish to become pregnant during the study
* Known chronic or severe infection or recent significant exposure to infections such as tuberculosis or endemic mycosis, untreated latent infections like tuberculosis, or a positive or indeterminate QuantiFERON test.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of imdusiran and durvalumab in NA suppressed CHB subjects | Up to 96 weeks
  • Number of participants with treatment emergent adverse events (TEAEs), immune related adverse events (irAEs), with discontinuations due to adverse events (AEs) and irAEs, with abnormal laboratory tests results, abnormal Vital signs, abnormal physical exam findings and abnormal electrocardiogram (ECG) readings

SECONDARY OUTCOMES:
To determine the effect of imdusiran and durvalumab on HBsAg | Up to 96 Weeks
  • Change in HBsAg levels from baseline during treatment and follow-up
To characterize the target engagement (TE) (pharmacodynamics [PD]) of durvalumab in CHB subjects over time | Up to 48 Weeks
  • Measurement of soluble immune marker levels in plasma at multiple timepoints
To determine the proportion of subjects who meet NA treatment discontinuation criteria at Week 48 | Up to Week 48
  • Proportion of subjects at Week 48 who are HBeAg negative and meet protocol defined ALT, HBV DNA and HBsAg values

CONTACTS AND LOCATIONS:
Locations (22):
- Georgia (2):
  - Infectious Diseases, AIDS and Clinical Immunology Research Center, Tbilisi
  - LLC "Neolab", Tbilisi
- Hong Kong (2):
  - Prince Of Wales Hospital - The Chinese University Of Hong Kong, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Poland (3):
  - Punkt Zdrowia Hlebowicz Jakubowski Lekarze Spółka Partnerska, Gdansk
  - ID Clinic Arkadiusz Pisula, Mysłowice
  - Punkt Zdrowia Hlebowicz Jakubowski Lekarze Spółka Partnerska, Wroclaw
- Arensia Exploratory Medicine Srl Romania in colaborare cu Institutul National de Boli Infectioase, Bucharest, Romania
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
- Taiwan (5):
  - Chia-yi Christian Hospital, Chia-Yi City
  - Kaohsiung Medical University Chung-ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Thailand (5):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - The Hiv Netherlands Australia Thailand Research Collaboration, Bangkok
  - Srinagarind Hospital, Khon Kaen
  - Naresuan University Hospital, Phitsanulok
- United Kingdom (2):
  - Imperial College Hospital, London
  - Royal London Hospital, London